CLINICAL TRIAL: NCT00885638
Title: Study of the Effect of Sitagliptin on the Hormonal Responses to Macronutrient Ingestion in Healthy Volunteers
Brief Title: Effects of Dipeptidyl Peptidase-4 (DPP-4) Inhibition on Hormonal Responses to Macronutrient Ingestion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Lund University Diabetes 001
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Healthy; Type 2 Diabetes
Keywords: GLP-1; Insulin secretion; Macronutrients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A placebo tablet is given before ingestion of macronutrients
  Interventions: Drug: placebo
- Sitagliptin (Active Comparator): Sitagliptin is given before ingestion of macronutrients
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — 100 mg sitagliptin before ingestion of macronutrient
  Other Names: Januvia
  Arms: Sitagliptin
Drug: placebo — A placebo tablet is given before ingestion of macronutrients
  Arms: Placebo

SUMMARY:
The regulation by DPP-4 inhibition after ingested of different individual macronutrients is not known. Therefore, this study examines the influence of ingestion of fat, protein, glucose or mixed meal on the concentrations of incretin hormones and insulin secretion with or without concomitant administration of a DPP-4 inhibitor (sitagliptin).

DETAILED DESCRIPTION:
Meal ingestion releases gut hormones which stimulate insulin secretion. A most important gut hormone is the incretin hormone glucagon-like peptide-1 (GLP-1). GLP-1 is rapidly degraded and inactivated after its release by the enzyme dipeptidyl peptidase-4 (DPP-4). Inhibition of DPP-4 therefore increases the concentration of active GLP-1 after meal ingestion, which augments insulin secretion. How this process is regulated after ingested of different individual macronutrients is not known. Therefore, this study examines the influence of ingestion of fat, protein, glucose or mixed meal on the concentrations of incretin hormones and insulin secretion with or without concomitant administration of a DPP-4 inhibitor (sitagliptin).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age 20-30 years
* BMI 20-30 kg/m2

Exclusion Criteria:

* Any disease
* Any medication

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Clinical Sciences Lund, Lund University, Lund, Sweden

REFERENCES:
- [Background] Carr RD, Larsen MO, Winzell MS, Jelic K, Lindgren O, Deacon CF, Ahren B. Incretin and islet hormonal responses to fat and protein ingestion in healthy men. Am J Physiol Endocrinol Metab. 2008 Oct;295(4):E779-84. doi: 10.1152/ajpendo.90233.2008. Epub 2008 Jul 8. PMID 18612044
- [Derived] Ohlsson L, Alsalim W, Carr RD, Tura A, Pacini G, Mari A, Ahren B. Glucose-lowering effect of the DPP-4 inhibitor sitagliptin after glucose and non-glucose macronutrient ingestion in non-diabetic subjects. Diabetes Obes Metab. 2013 Jun;15(6):531-7. doi: 10.1111/dom.12062. Epub 2013 Feb 7. PMID 23331498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed during 2011 to Lund University
Groups:
- Placebo First, Then Sitagliptin; Sitagliptin First, Then Placebo: First intervention 1 day, washout 14 days, second intervention 1 day
Period: Overall Study
Arm/Group | Placebo First, Then Sitagliptin | Sitagliptin First, Then Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Placebo first, then sitagliptin or sitagliptin first, then placebo
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  Sweden | 12

OUTCOME MEASURES:

1. Primary Outcome: Glucagon-like Peptide-1 Secretion After Meal Ingestion
Description: Plasma GLP-1 levels will be measured during 300 min after meal ingestion for estimation of GLP-1 secretion
Time Frame: 300 min
Population: Completer population
Measure: Mean (Standard Error); unit: nmol/l/min
Groups:
- Placebo: Placebo first, then sitagliptin or sitagliptin first, then placebo; this is the result for placebo
- Sitagliptin: Placebo first, then sitagliptin or sitagliptin first, then placebo; this is the result for sitagliptin
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 12 | 12
nmol/l/min | 0.82 (0.11) | 1.24 (0.13)

2. Secondary Outcome: Insulin Secretion After Ingestion of Meal
Description: Plasma insulin levels will be measured during 300 min after meal ingestion to estimation of insulin secretion
Time Frame: 300 min
Population: Completer population
Measure: Mean (Standard Error); unit: mol/l/min
Groups:
- Placebo: A placebo tablet is given before ingestion of meal
- Sitagliptin: Sitagliptin is given before ingestion of meal
Arm/Group | Placebo | Sitagliptin
Number analyzed (Participants) | 12 | 12
mol/l/min | 29.6 (2.8) | 24.7 (2.2)

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No